CLINICAL TRIAL: NCT00552877
Title: Randomized Clinical Comparison of the Xience V and the Cypher Coronary Stents in Non-selected Patients With Coronary Heart Disease
Brief Title: The SOURT OUT IV TRIAL
Acronym: SORT OUT IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Per Thayssen, Odense University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SOIV-20070043
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Ischemic Heart Disease; Coronary Atherosclerosis; Percutaneous Coronary Intervention
Keywords: PCI; Drug-eluting stent
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Cypher Select plus stent
  Interventions: Device: Percutaneous coronary intervention (Xience V stent)
- 2 (Active Comparator): Xience V stent
  Interventions: Device: Percutaneous coronary intervention (Xience V stent)

INTERVENTIONS:
Device: Percutaneous coronary intervention (Xience V stent) — Cypher Select plus coronary stent Xience V coronary stent
  Other Names: Cypher Select plus coronary stent; Xience V coronary stent

SUMMARY:
In a randomized study the Xience V coroary artery stent may be non inferior to the Cypher Select+ coronary stents in the treatment of unselected patients with coronary artery disease.

DETAILED DESCRIPTION:
2 Purpose In a randomized study to compare the Cypher Select+ and the Xience V coronary stents in the treatment of unselected patients with coronary artery disease.

2.1 Primary objective In a randomized study to compare the Xience V and the Cypher Select+ coronary stents by assessing SAFETY (cardiac death, myocardial infarction and/or stent thrombosis) and EFFICACY (target vessel revascularization) after 9 months.

2.2 Secondary objective To compare device success rate, procedure success rate and complication rate during hospitalization, after 1 month and after 9 months and the incidence of late stent thrombosis after 12, 24 and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with one or more drug eluting stents in the coronary arteries at one of the 5 heart centres in Denmark (Gentofte, Rigshospitalet, Odense, Skejby, Aalborg) can be included in the study.

Exclusion Criteria:

* The patient will not participate
* The patient participates in other randomised stent studies
* Expected survival < 1 year
* Allergy to Aspirin, Clopidogrel or Ticlopidine
* Allergy to Sirolimus or ABT-578

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2678 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
SAFETY (cardiac death, myocardial infarction and/or stent thrombosis) EFFICACY (target vessel revascularization) | 9 months, 1 year, 2 years, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Per Thayssen, MD DMSci, Principal Investigator — Odense University Hospital, Dept. of Cardiology
Locations (1):
- Odense University Hospital, Dept. of Cardiology, Odense, Denmark

REFERENCES:
- [Derived] Jensen LO, Thayssen P, Christiansen EH, Maeng M, Ravkilde J, Hansen KN, Hansen HS, Krusell L, Kaltoft A, Tilsted HH, Berencsi K, Junker A, Lassen JF; SORT OUT IV Investigators. Safety and Efficacy of Everolimus- Versus Sirolimus-Eluting Stents: 5-Year Results From SORT OUT IV. J Am Coll Cardiol. 2016 Feb 23;67(7):751-62. doi: 10.1016/j.jacc.2015.11.051. PMID 26892409
- [Derived] Jensen LO, Thayssen P, Maeng M, Christiansen EH, Ravkilde J, Hansen KN, Kaltoft A, Tilsted HH, Madsen M, Lassen JF; Scandinavian Organization for Randomized Trials With Clinical Outcome SORT OUT IV Investigators. Three-year outcomes after revascularization with everolimus- and sirolimus-eluting stents from the SORT OUT IV trial. JACC Cardiovasc Interv. 2014 Aug;7(8):840-8. doi: 10.1016/j.jcin.2014.02.014. Epub 2014 Jul 30. PMID 25086842
- [Derived] Antonsen L, Thayssen P, Hansen HS, Maeng M, Tilsted HH, Botker HE, Ravkilde J, Madsen M, Sorensen HT, Thuesen L, Lassen JF, Jensen LO. Outcomes after revascularisation with everolimus- and sirolimus-eluting stents in patients with acute coronary syndromes and stable angina pectoris: a substudy of the SORT OUT IV trial. EuroIntervention. 2014 Jun;10(2):212-23. doi: 10.4244/EIJV10I2A35. PMID 23838425
- [Derived] Jensen LO, Thayssen P, Christiansen EH, Tilsted HH, Maeng M, Hansen KN, Kaltoft A, Hansen HS, Botker HE, Krusell LR, Ravkilde J, Madsen M, Thuesen L, Lassen JF; SORT OUT IV Investigators. 2-year patient-related versus stent-related outcomes: the SORT OUT IV (Scandinavian Organization for Randomized Trials With Clinical Outcome IV) Trial. J Am Coll Cardiol. 2012 Sep 25;60(13):1140-7. doi: 10.1016/j.jacc.2012.07.004. Epub 2012 Sep 5. PMID 22958957
- [Derived] Jensen LO, Thayssen P, Hansen HS, Christiansen EH, Tilsted HH, Krusell LR, Villadsen AB, Junker A, Hansen KN, Kaltoft A, Maeng M, Pedersen KE, Kristensen SD, Botker HE, Ravkilde J, Sanchez R, Aaroe J, Madsen M, Sorensen HT, Thuesen L, Lassen JF; Scandinavian Organization for Randomized Trials With Clinical Outcome IV (SORT OUT IV) Investigators. Randomized comparison of everolimus-eluting and sirolimus-eluting stents in patients treated with percutaneous coronary intervention: the Scandinavian Organization for Randomized Trials with Clinical Outcome IV (SORT OUT IV). Circulation. 2012 Mar 13;125(10):1246-55. doi: 10.1161/CIRCULATIONAHA.111.063644. Epub 2012 Feb 3. PMID 22308301
- [Derived] Jensen LO, Thayssen P, Tilsted HH, Ravkilde J, Junker A, Hansen HS, Hansen KN, Pedersen KE, Sorensen HT, Thuesen L, Lassen JF; Scandinavian Organization for Randomized Trials with Clinical Outcome SORT OUT IV investigators. Rationale and design of a randomized clinical comparison of everolimus-eluting (Xience v/Promus) and sirolimus-eluting (cypher select+) coronary stents in unselected patients with coronary heart disease. Cardiology. 2010;116(2):73-8. doi: 10.1159/000315136. Epub 2010 Jun 3. PMID 20523042